CLINICAL TRIAL: NCT00745420
Title: Unrelated Donor Reduced Intensity Bone Marrow Transplant for Children With Severe Sickle Cell Disease (BMT CTN #0601)
Brief Title: Evaluating the Safety and Effectiveness of Bone Marrow Transplants in Children With Sickle Cell Disease (BMT CTN 0601)
Acronym: SCURT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other); Sickle Cell Disease Clinical Research Network (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0601; U01HL069294 (NIH); 5U24CA076518 (NIH)
Record Dates: First submitted 2008-08-29; First posted 2008-09-03 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hematopoietic Stem Cell Transplantation; Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hematopoietic Stem Cell Transplantation (Experimental): Bone Marrow Transplant with GVHD Prophylaxis Regimen
  Interventions: Biological: Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Biological: Hematopoietic Stem Cell Transplantation — The stem cell transplant preparative regimen is listed below. Day 0 is the day of the transplant. The - sign is the number of days before and the + sign is the number of days after the transplant.
  * Alemtuzumab: Children weighing 10 kg or more will receive 10 mg, 15 mg, and 20 mg intravenously (IV) on Days -21, -20, and -19, respectively
  * Fludarabine: 30 mg/m^2/day IV on Days -8 through -4
  * Melphalan: 140 mg/m^2 IV on Day -3
  * Rest on Days -2 and -1
  * Transplant occurs on Day 0
  * GVHD prophylaxis: Tacrolimus or cyclosporine beginning Day -3, methotrexate (7.5 mg/m2/day) Day 1, 3 and 6 and methylprednisolone/prednisone on Day +7 to +28 followed by a taper if there is no GVHD
  Other Names: Bone Marrow Transplant

SUMMARY:
Sickle cell disease (SCD), also known as sickle cell anemia, is an inherited blood disease that can cause organ damage, stroke, and intense pain episodes. A blood stem cell transplant is a treatment option for someone with a severe form of the disease. Prior to undergoing a transplant, people typically receive a conditioning regimen of high doses of chemotherapy and other medications to prepare the body to accept the transplant. A conditioning regimen that uses lower doses of chemotherapy and medications may be safer for transplant recipients. This study will evaluate the safety and effectiveness of blood stem cell transplants, using bone marrow from unrelated donors, in children with severe SCD who receive a reduced intensity conditioning regimen prior to the transplant.

DETAILED DESCRIPTION:
SCD is an inherited blood disorder. Symptoms include anemia, infections, organ damage, and intense episodes of pain, also called "sickle cell crises." SCD is caused by an abnormal type of hemoglobin, which is a protein inside red blood cells that carries oxygen to vital organs, such as the brain, heart, lungs, and kidneys. Defective hemoglobin damages red blood cells. The damaged cells, in turn, can block blood flow in vessels and block oxygen and nutrients from reaching organs. For people with severe forms of SCD, one treatment option is a bone marrow transplant, which may correct the abnormal blood cell production problem. In most cases, bone marrow transplants are performed in people who have a healthy sibling with the same tissue type. If people do not have a sibling with the same tissue type, it is possible for them to receive a blood stem cell transplant from an unrelated donor through bone marrow transplant .

Traditionally, people with SCD who are undergoing a bone marrow transplant receive high doses of chemotherapy and medications before the transplant as part of the conditioning regimen to prepare their immune system to accept the donor cells. Participants will experience fewer side effects with a reduced intensity conditioning regimen than with a more intense conditioning regimen. The purpose of this study is to determine the safety and effectiveness of blood stem cell transplants, using bone marrow from unrelated donors, in children with severe SCD who receive a reduced intensity conditioning regimen before the transplant. Specifically, researchers will evaluate whether the reduced intensity conditioning regimen is successful in allowing donor cells to settle and grow successfully, in preventing the production of SCD-damaged red blood cells, and in limiting SCD-related organ damage.

This study will enroll children with severe SCD who lack a sibling with the same tissue type who can serve as their donor. Participants will attend a study visit prior to the transplant to undergo a blood collection, neurocognitive testing to measure learning and brain function, and magnetic resonance angiogram (MRA) and magnetic resonance imaging (MRI) scans. Questionnaires to assess quality of life will also be completed. Twenty-two days before the transplant, participants will begin receiving a reduced intensity conditioning regimen of chemotherapy and medications to prepare them for the transplant. Eight days before the transplant, participants will be admitted to the hospital and will continue the conditioning regimen. Participants will then receive the bone marrow transplant. After the transplant, participants will receive immunosuppression medications for at least 6 months to prevent graft-versus-host disease (GVHD), which may occur if the immune cells from the donated bone marrow attacks the body of the recipient. One week after the transplant, participants will receive granulocyte-colony-stimulating factor (G-CSF), which is a natural protein that increases the white blood cell count and helps protect the body against infections. Participants will receive G-CSF until their white blood cell level is normal again. Participants will remain in the hospital and be closely monitored for signs of infection or other complications until study researchers feel it is safe for them to return home.

After leaving the hospital, participants will attend study visits weekly during Weeks 1 to 8, at Day 60, weekly during Weeks 9 to 14, at Day 100, at Month 6, and at Years 1 and 2. At all study visits, a blood collection, medical history review, and physical exam will occur. In addition, at Day 100, Month 6, and Years 1 and 2, questionnaires to assess quality of life will be completed. At select visits the following procedures will also occur: lung function testing, heart function testing, MRA and MRI scans, and neurocognitive testing.

ELIGIBILITY:
Inclusion Criteria:

* SCD (genotype hemoglobin SS disease [Hb SS], genotype hemoglobin SC disease [HbSC],sickle ß°[Sß°] thalassemia, or sickle ß^+[Sß^+]thalassemia) with one or more of the following:

  1. Patients must have symptomatic SCD (genotype Hb SS, Hb SC, Sß° thalassemia or Sß+ thalassemia), AND have 1 or more of the following clinical complications:(i) Clinically significant neurologic event (stroke) or any neurologic deficit lasting more than 24 hours that is accompanied by an infarct on cerebral MRI; OR (ii) patients who have a Transcranial Doppler (TCD) velocity that exceeds 200 cm/sec by the non-imaging technique (or TCD measurement greater than 185 cm/sec by the imaging technique) measured at a minimum of 2 separate occasions one month or more apart; OR,
  2. Minimum of two episodes of acute chest syndrome in the 2 years before study entry, defined as new pulmonary alveolar consolidation involving at least one complete lung segment (associated with acute symptoms including fever, chest pain, tachypnea, wheezing, rales, or cough that is not attributed to asthma or bronchiolitis) despite adequate supportive care measures
  3. History of 3 or more severe pain events per year in the 2 years before study entry
* Lansky/Karnofsky performance score greater than or equal to 40
* Patients must have an unrelated adult bone marrow donor who is Human Leukocyte Antigen (HLA)-matched at 8 of 8 HLA-A, -B, -C and -DRB1 at high resolution using DNA-based typing.
* Patients with adequate physical function: a)Cardiac: Left ventricular ejection fraction (LVEF) greater than 40%, or LV shortening fraction greater than 26%; b) Pulmonary: Pulse oxymetry with a baseline O2 saturation of greater than or equal to 85% is required for all patients, Carbon Monoxide Diffusing Capacity (DLCO) greater than 40% (corrected for hemoglobin) for patients in whom pulmonary function testing can be performed; c) Renal: Serum creatinine less than or equal to 1.5 x upper limit of normal for age and glomerular filtration rate (GFR) greater than 100 mL/min/1.73 m. For patients older than or equal to 16 years of age, GFR should be greater than 70 mL/min/1.73 m^2; d) Hepatic: Serum conjugated (direct) bilirubin less than 2x upper limit of normal for age as per local laboratory; alanine transaminase (ALT) and aspartate transaminase (AST) less than 5 times upper limit of normal as per local laboratory.
* If the patient has been receiving chronic transfusion therapy for more than or equal to 1 year AND has clinical evidence of iron overload (serum ferritin level of greater than 1000 ng/ml), a liver biopsy shall be obtained within 90 days of starting conditioning therapy (alemtuzumab). Histologic exam of the liver must document absence of bridging fibrosis or cirrhosis of the liver. In other cases, a liver biopsy is optional.
* Hemoglobin S (Hb S) level less than or equal to 45%, seven days prior to initiation of alemtuzumab

Exclusion Criteria:

* Evidence of uncontrolled bacterial, viral or fungal infections (currently taking medication and progression of clinical symptoms) within 1 month prior to starting the conditioning regimen. Patients with fever or suspected minor infection should await resolution of symptoms before starting the conditioning regimen
* Pregnant or breastfeeding
* Patients with 8/8 HLA-matched family donors able to donate
* Seropositivity for HIV
* Prior allogeneic marrow or stem cell transplant
* Iron chelation must be discontinued more than or equal to 48 hours before initiating the conditioning regimen
* Hydroxyurea (if receiving this therapy) must be discontinued more than or equal to 48 hours before initiating the conditioning regimen

Ages: 3 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2015-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital of New Orleans/LSUMC CCOP, New Orleans, Louisiana
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Washington University, St. Louis Children's Hospital, St Louis, Missouri
  - Cohen Children's Hospital, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine/The Methodist Hospital, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076
- [Result] Shenoy S, Eapen M, Panepinto JA, Logan BR, Wu J, Abraham A, Brochstein J, Chaudhury S, Godder K, Haight AE, Kasow KA, Leung K, Andreansky M, Bhatia M, Dalal J, Haines H, Jaroscak J, Lazarus HM, Levine JE, Krishnamurti L, Margolis D, Megason GC, Yu LC, Pulsipher MA, Gersten I, DiFronzo N, Horowitz MM, Walters MC, Kamani N. A trial of unrelated donor marrow transplantation for children with severe sickle cell disease. Blood. 2016 Nov 24;128(21):2561-2567. doi: 10.1182/blood-2016-05-715870. Epub 2016 Sep 13. PMID 27625358
- [Derived] Martens MJ, Logan BR. Statistical rules for safety monitoring in clinical trials. Clin Trials. 2024 Apr;21(2):152-161. doi: 10.1177/17407745231203391. Epub 2023 Oct 25. PMID 37877375
- [Derived] Leonard A, Furstenau D, Abraham A, Darbari DS, Nickel RS, Limerick E, Fitzhugh C, Hsieh M, Tisdale JF. Reduction in vaso-occlusive events following stem cell transplantation in patients with sickle cell disease. Blood Adv. 2023 Jan 24;7(2):227-234. doi: 10.1182/bloodadvances.2022008137. PMID 36240296

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between August 2008 and April 2014 from 19 different transplant centers.
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplantation
Started | 30
Completed | 29
Not Completed | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 14 [6 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 26
  Hispanic or Latino | 3
Indications for Transplant [Count of Participants; unit: Participants] — Some patients had more than 1 indication
  Participants
    Stroke | 12
    Trans cranial doppler velocity > 200cm/s | 2
    Acute chest syndrome | 4
    Vaso-occlusive pain crisis | 12
Chronic Blood Transfusion Prior to Transplant [Count of Participants; unit: Participants] | 14
Karnofsky Performance Score [Count of Participants; unit: Participants] — Assesses patient self-perceived global quality of life and functioning on a scale of 0 - 100; where 100 equals normal quality of life with no evidence of disease, 90 equals ability to carry on normal activity with minor signs/symptoms of disease, 80 equals normal activity with effort and some signs/symptoms of disease, and 70 equals ability to care for oneself but unable to carry on normal activity or to do active work.
  Participants
    100 | 17
    90 | 9
    80 | 2
    70 | 1
Cytomegalovirus (CMV) Status [Count of Participants; unit: Participants]
  CMV - donor and recipient | 8
  CMV + donor and recipient | 9
  CMV - donor and CMV + recipient | 3
  CMV + donor and CMV - recipient | 9
Donor Blood Type Match [Count of Participants; unit: Participants]
  ABO Blood group matched | 15
  ABO Blood group major mismatch | 9
  ABO Blood group minor mismatch | 5
Donor Gender Match [Count of Participants; unit: Participants]
  Gender matched transplants | 15
  Female donor, male recipient | 7
  Male donor, female recipient | 7
Donor Age [Median (Full Range); unit: years] | 35 [21 to 55]
Donor Race/Ethnicity [Count of Participants; unit: Participants]
  Caucasian | 11
  Black or African American | 11
  Multiracial | 5
  Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Event-Free Survival (EFS)
Description: EFS is defined as percentage of participants that have not had an event. Primary or secondary graft rejection, disease recurrence, or death will count as events for this endpoint.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 29
percentage of participants
  1 year | 76 [56 to 88]
  2 years | 69 [48 to 82]

2. Secondary Outcome: Percentage of Participants With Overall Survival (OS)
Description: OS is defined as the percentage of participants that have not died.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 29
percentage of participants
  1 year | 86 [67 to 95]
  2 years | 79 [59 to 90]

3. Secondary Outcome: Neutrophil and Platelet Recovery
Description: Time to neutrophil recovery is defined as the time of the first of three measurements on consecutive days where the patient has an absolute neutrophil count of >= 500/uL following conditioning regimen induced nadir. Time to platelet recovery is defined as the time of the first of three measurements on consecutive days where the patient has achieved a platelet count > 50,000/uL and is platelet transfusion independent for a minimum of seven days following conditioning regimen induced nadir.
Time Frame: Up to 100 days
Measure: Median (Full Range); unit: days
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 29
days
  Neutrophil Recovery | 12 [6 to 16]
  Platelet Recovery | 24 [7 to 90]

4. Secondary Outcome: Graft Rejection
Description: Primary graft rejection is defined as the presence of less than 20% donor cells as assessed by peripheral blood or bone marrow chimerism assays on or after Day 42. Secondary graft rejection is defined as the presence of less than 20% donor derived hematopoietic cells in peripheral blood or bone marrow that occurs after prior evidence of 20% or greater donor cells.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 29
Participants
  Primary Graft Rejection | 2
  Secondary Graft Rejection | 1

5. Secondary Outcome: Percentage of Participants With Acute Graft-vs-Host-Disease (GVHD)
Description: Acute GVHD is graded according to the scoring system proposed by Przepiorka et al.1995:
  Skin stage:
  0: No rash
  1. Rash <25% of body surface area
  2. Rash on 25-50% of body surface area
  3. Rash on > 50% of body surface area
  4. Generalized erythroderma with bullous formation
  Liver stage (based on bilirubin level)*:
  0: <2 mg/dL
  1. 2-3 mg/dL
  2. 3.01-6 mg/dL
  3. 6.01-15.0 mg/dL
  4. >15 mg/dL
  GI stage*:
  0: No diarrhea or diarrhea <500 mL/day
  1. Diarrhea 500-999 mL/day or persistent nausea with histologic evidence of GVHD
  2. Diarrhea 1000-1499 mL/day
  3. Diarrhea >1500 mL/day
  4. Severe abdominal pain with or without ileus * If multiple etiologies are listed for liver or GI, the organ system is downstaged by 1.
  GVHD grade:
  0: All organ stages 0 or GVHD not listed as an etiology I: Skin stage 1-2 and liver and GI stage 0 II: Skin stage 3 or liver or GI stage 1 III: Liver stage 2-3 or GI stage 2-4 IV: Skin or liver stage 4
Time Frame: 100 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 29
percentage of participants
  Grade II-IV Acute GVHD | 28 [13 to 45]
  Grade III-IV Acute GVHD | 17 [6 to 33]

6. Secondary Outcome: Percentage of Participants With Chronic GVHD
Description: Chronic GVHD is defined per NIH 2005 Consensus Criteria.
Time Frame: 1 year post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 29
percentage of participants | 62 [41 to 77]

7. Secondary Outcome: Number of Participants With Chronic GVHD by Severity
Description: Chronic GVHD severity is defined per NIH 2005 Consensus Criteria.
Time Frame: 1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 29
Participants
  None | 10
  Mild | 6
  Moderate | 8
  Severe | 5

8. Secondary Outcome: Percentage of Participants With Posterior Reversible Encephalopathy Syndrome (PRES)
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 29
percentage of participants | 34 [18 to 52]

9. Secondary Outcome: Change From Baseline to Day 100 in Participant Reported Health-Related Quality of Life (HRQL)
Description: HRQL will be assessed using the Self-Esteem, General Health Perception, and Change in Health subscales of the Child Health Questionnaire (CHQ Child Form 87). The changes in participant reported scores on these HRQL subscales from a pre-transplant baseline assessment to day 100 post-transplant will be evaluated. Each subscale is scored is scored in the range 0-100, with higher scores indicating better health and well-being. Therefore, a negative mean change in score denotes worsening HRQL score and positive mean change in score denotes an improved HRQL score over time.
Time Frame: 100 days post-transplant
Population: Participants age 10 years or older that returned the HRQL surveys
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 18
units on a scale
  Self esteem score | -0.59 (4.51)
  General health perception score | -1.90 (4.29)
  Change in health score | 0.33 (0.45)

10. Secondary Outcome: Change From Baseline to Day 100 in Parent Proxy Reported Health-Related Quality of Life (HRQL)
Description: HRQL will be assessed using the Self-Esteem, General Health Perception, and Change in Health subscales of the Child Health Questionnaire (CHQ Child Form 87). The changes in parent proxy reported scores on these HRQL subscales from a pre-transplant baseline assessment to day 100 post-transplant will be evaluated. Each subscale is scored is scored in the range 0-100, with higher scores indicating better health and well-being. Therefore, a negative mean change in score denotes worsening HRQL score and positive mean change in score denotes an improved HRQL score over time.
Time Frame: 100 days post-transplant
Population: Parent proxies of participants that returned the HRQL surveys
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 21
units on a scale
  Self esteem scale score | -15.12 (4.89)
  General health perception score | 11.13 (2.51)
  Change in health score | 0.90 (0.38)

11. Secondary Outcome: Change From Baseline to Day 180 in Participant Reported Health-Related Quality of Life (HRQL)
Description: HRQL will be assessed using the Self-Esteem, General Health Perception, and Change in Health subscales of the Child Health Questionnaire (CHQ Child Form 87). The changes in participant reported scores on these HRQL subscales from a pre-transplant baseline assessment to day 180 post-transplant will be evaluated. Each subscale is scored is scored in the range 0-100, with higher scores indicating better health and well-being. Therefore, a negative mean change in score denotes worsening HRQL score and positive mean change in score denotes an improved HRQL score over time.
Time Frame: 180 days post-transplant
Population: Participants age 10 years or older that returned the HRQL surveys
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 16
units on a scale
  Self esteem scale score | -4.33 (5.87)
  General health perception score | -6.69 (4.99)
  Change in health score | 0.19 (0.52)

12. Secondary Outcome: Change From Baseline to Day 180 in Parent Proxy Reported Health-Related Quality of Life (HRQL)
Description: HRQL will be assessed using the Self-Esteem, General Health Perception, and Change in Health subscales of the Child Health Questionnaire (CHQ Child Form 87). The changes in parent proxy reported scores on these HRQL subscales from a pre-transplant baseline assessment to day 180 post-transplant will be evaluated. Each subscale is scored is scored in the range 0-100, with higher scores indicating better health and well-being. Therefore, a negative mean change in score denotes worsening HRQL score and positive mean change in score denotes an improved HRQL score over time.
Time Frame: 180 days post-transplant
Population: Parent proxies of participants that returned the HRQL surveys
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 20
units on a scale
  Self esteem scale score | -11.46 (6.28)
  General health perception score | 7.63 (3.31)
  Change in health score | 1.15 (0.36)

13. Secondary Outcome: Change From Baseline to 1 Year in Participant Reported Health-Related Quality of Life (HRQL)
Description: HRQL will be assessed using the Self-Esteem, General Health Perception, and Change in Health subscales of the Child Health Questionnaire (CHQ Child Form 87). The changes in participant reported scores on these HRQL subscales from a pre-transplant baseline assessment to 1 year post-transplant will be evaluated. Each subscale is scored is scored in the range 0-100, with higher scores indicating better health and well-being. Therefore, a negative mean change in score denotes worsening HRQL score and positive mean change in score denotes an improved HRQL score over time.
Time Frame: 1 year post-transplant
Population: Participants age 10 years or older that returned the HRQL surveys
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 13
units on a scale
  Self esteem scale score | 4.97 (5.33)
  General health perception score | 6.99 (6.35)
  Change in health score | 1.46 (0.35)

14. Secondary Outcome: Change From Baseline to 1 Year in Parent Proxy Reported Health-Related Quality of Life (HRQL)
Description: HRQL will be assessed using the Self-Esteem, General Health Perception, and Change in Health subscales of the Child Health Questionnaire (CHQ Child Form 87). The changes in parent proxy reported scores on these HRQL subscales from a pre-transplant baseline assessment to 1 year post-transplant will be evaluated. Each subscale is scored is scored in the range 0-100, with higher scores indicating better health and well-being. Therefore, a negative mean change in score denotes worsening HRQL score and positive mean change in score denotes an improved HRQL score over time.
Time Frame: 1 year post-transplant
Population: Parent proxies of participants that returned the HRQL surveys
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 15
units on a scale
  Self esteem scale score | -3.61 (6.66)
  General health perception score | 8.89 (5.27)
  Change in health score | 1.53 (0.48)

ADVERSE EVENTS:
Time Frame: 2 years post-transplant
Description: Serious Adverse Events (AE) are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event. Only unexpected grades 3-5 adverse events were required to be reported through the AE system per protocol.
Arm/Group | Hematopoietic Stem Cell Transplantation
Serious Adverse Events (participants affected / at risk) | 21/29
Other Adverse Events (participants affected / at risk) | 2/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=29)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=29)
Seizure (Nervous system disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2014-06-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT00745420/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2015-05-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT00745420/SAP_001.pdf